CLINICAL TRIAL: NCT06313489
Title: Rupture of Extensor Pollicis Longus Tendon After Fracture of the Distal Radius, Study of Muscle and Tendon Pathology
Brief Title: Rupture of Thumb's Long Extensor Tendon After Fracture of the Distal Radius, Study of Muscle and Tendon Pathology
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Anders Bjorkman, Professor, Göteborg University
Other Study IDs: 282151
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Distal Radius Fractures; Tendon Injury - Hand; Pathology
Keywords: Extensor pollicis longus rupture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Specimens of EPL muscle and tendon in cases of tendon rupture after fractures of the distal radius
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with ruptures of Extensor pollicis longus tendon after distal radial fracture: Patients planned for intervention according to the clinical practice. We planned to include all patients that would be treated in out department.
  Interventions: Procedure: Biopsy of EPL tendon and muscle during the operation

INTERVENTIONS:
Procedure: Biopsy of EPL tendon and muscle during the operation — Biopsy of EPL tendon and muscle

SUMMARY:
Fractures of the wrist (fractures of the distal radius) are one of the most common fractures with almost 60 000 injuries per year in Sweden. One known complication following these fractures is that the long extensor tendon of the thumb ruptures (extensor pollicis longus tendon, EPL tendon). This leads to disability to stretch the thumb in order to grip bigger objects. Earlier studies show that the tendon ruptures in about 3-5% of all wrist fractures. These ruptures occur some weeks to months after the fracture.

There are different theories about the cause of the rupture. One theory is that the fracture creates a bleeding in the tight area that the tendon lies, leading to high pressure and therefore low blood supply to the tendon. Another theory is that the tendon comes in contact with some sharp bonny fragments in this area that injures the tendon when it moves.

Such tendon ruptures need almost always some type of surgical intervention in order to reconstruct the function of the thumb. A common problem is that the quality of the tendon is insufficient for just suturing it. Another problem is that the muscle becomes stiff after the rupture. However, there is no objective method to determine how stiff the muscle is.

The most common treatment option is the transfer of one of the two extensor tendons of the index finger to the thumb, a so-called extensor indicis proprius to extensor pollicis longus transfer. The motivation behind this operation is that the muscle of EPL is so stiff that cannot be used to lift the thumb. However, there is no consensus about the time period after which the EPL muscle can be used to reconstruct the function of thumb.

The study aims to investigate the microscopical changes in the muscle and tendon of EPL after such a rupture. Better knowledge of these factors could lead to better understanding of the treatment options.

The investigators plan to include in the study all patients that would get operated for an EPL tendon rupture after a fracture of the distal radius at the institution the study is conducted. After oral and written information to the patient and written consent the investigators will take some samples from the ruptured tendon and muscle for microscopical analysis.

DETAILED DESCRIPTION:
Ruptures of extensor pollicis longus (EPL) tendon are a known complication of fractures of the distal radius. The study plan is to conduct a prospective histopathological study of the EPL muscle and tendon on patients operated for ruptures of EPL after fractures of the distal radius.

The standard treatment at the institution the study is conducted is a tendon transfer of extensor indicis proprius to EPL. Under this operation the investigators plan to take tissue biopsies from the distal part of the muscle and the ruptured tendon and conduct a histopathological analysis.

Participants received oral and written information and left a written consent. The participants were assessed for sex, age, relevant medication and prior surgical interventions in the hand and wrist. Epidemiological data for the fracture time, classification and treatment is documented as well epidemiological data for the tendon rupture.

The histopathological analysis is conducted by one researcher in the group, expert in muscle pathology.

ELIGIBILITY:
Inclusion Criteria:

* a clinically diagnosed EPL rupture after a fracture of the distal radius

Exclusion Criteria:

* Inability to read and understand Swedish
* Mental illness leading to inability to understand the study procedure or rehabilitation training.
* Active drug use.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with rupture of EPL after fractures of the distal radius at Sahlgrenska University Hospital at the department of Orthopaedic Traumatology and at the department of Hand surgery. The patients should be eligible for surgical reconstruction of EPL according to the clinical practise.
  Sahlgrenska University Hospital covers the metropolitan area of Gothenburg with a population of 1 million. Furthermore Sahlgrenska University Hospital is referral hospital for the greater region covering a population of about 2 millions.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Histopathological analysis of the EPL muscle | Analysis within 8 weeks from sampling
  Histochemical analyses, Muscle fiber typing,immunostainings brightfield microscopy. Selected specimens were also immuno-stained with inflammatory cell markers

SECONDARY OUTCOMES:
Histopathological analysis of the EPL tendon | Analysis within 8 weeks from sampling
  immunostainings brightfield microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Anders Björkman, Prof., Principal Investigator — Sahlgrenska University Hospital, University of Gothenburg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Västra Götaland County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarigiannis CN, Ullman M, Andreasson I, Oldfors A, Bjorkman A. Inflammatory and degenerative changes in the extensor pollicis longus muscle and tendon following ruptures caused by distal radius fractures. BMC Musculoskelet Disord. 2025 Jan 3;26(1):10. doi: 10.1186/s12891-024-08212-4. PMID 39754134